CLINICAL TRIAL: NCT01241682
Title: Dendritic Cell-based Immunotherapy Combined With Low-dose Cyclophosphamide in Patients With Malignant Mesothelioma
Acronym: PMR-MM-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, joost hegmans, Dr., Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL24050.000.08
Record Dates: First submitted 2010-06-01; First posted 2010-11-16 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Malignant (Pleural) Mesothelioma
Keywords: Mesothelioma; Dendritic cells; Cyclophosphamide; Tumor lysate-loaded; Immunotherapy
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC immunotherapy + CTX (Experimental): Patients with mesothelioma who are fit enough to be treated with chemotherapy and enough tumor material was available are asked for participation in this study. After 4 cycles of Alimta chemotherapy, a leukapheresis is performed of which the monocytes are used for differentiation to DCs using different cytokines. The procedure to grow DCs in vitro and pulse them with tumor lysate is performed according to our earlier performed phase I study that was approved by our local ethics committee. Three doses of properly pulsed autologous DCs (MesoCancerVac) are then re-injected every two weeks. Patients will be treated with a low dose of CTX for seven day in a row the week before the 1st vaccination, the weeks in between the 2nd, and for one week after the 3rd vaccination.
  Interventions: Biological: DC + CTX

INTERVENTIONS:
Biological: DC + CTX — 3x 50x10e6 DC + cyclophosphamide
  Other Names: Endoxan

SUMMARY:
Earlier the investigators determined the safety and feasibility of tumor lysate-pulsed dendritic cells as therapeutic adjuvants in mesothelioma patients. Because pre-clinical data in mice had shown that better results were obtained when regulatory T cells were depleted using low-dosis of cyclophosphamide, ten patients who responded on chemotherapy are selected for DC-treatment in combination with Endoxan.

DETAILED DESCRIPTION:
Currently there is no satisfactory low-toxicity treatment for patients with mesothelioma (MM). Based on studies in other types of cancer in humans where beneficial effects were obtained, and based on our pre-clinical data in a mouse model for MM, led to the introduction of DC-immunotherapy for human MM in 2005. A beneficial effect of immunotherapy in MM patients without major side effects was found, however, research has shown that DC immunotherapy might be further improved. The objectives of the here proposed phase study are:

* To define the safety and toxicity of low dose CTX in combination with MesoCancerVac in patients with MM.
* To determine if vaccination with low dose CTX in combination with MesoCancerVac results in a detectable immune response by skin DTH reactions on MM crude antigen and KLH and by in vitro laboratory analysis.
* To observe and document anti-cancer activity by laboratory evaluation (e.g. decrease in Tregs, increase in CTLs using 51Cr release and IFN-gamma ELISPOT)
* To observe and document anti-cancer activity by clinical evaluation (e.g. CT scan)

ELIGIBILITY:
Inclusion criteria:

* Patients with clinically and histological or cytological confirmed newly diagnosed MM, that can be measured in two dimensions by a radiologic imaging study.
* Patients must be at least 18 years old and must be able to give written informed consent.
* Patients must be ambulatory (Karnofsky scale > 70, or WHO-ECOG performance status 0,1, or 2) and in stable medical condition. The expected survival must be at least 4 months.
* Patients must have normal organ function and adequate bone marrow reserve: absolute neutrophil count > 1.5 x 109/l, platelet count > 100 x 109/l, and Hb > 6.0 mmol/l.
* Positive DTH skin test (induration > 2mm after 48 hrs) against at least one positive control antigen tetanus toxoid.
* Stable disease or response after chemotherapy.
* Availability of sufficient tumor material of the patient.
* Ability to return to the Erasmus MC for adequate follow-up as required by this protocol.
* Able to tolerate oral therapy
* No impairment of gastrointestinal (GI) function or GI disease that may affect or alter absorption of CTX (e.g., mal-absorption syndrome, history of total gastrectomy/significant small bowel resection)
* No history of allergic reactions (≥ grade 3 or 4) to compounds of similar chemical or biologic composition to CTX (i.e., alkylating agents)
* No known intolerance or hypersensitivity reaction to CTX

Exclusion criteria:

* Conditions that make the patient unfit for chemotherapy or progressive disease after 4 cycles of chemotherapy.
* Pleurodesis at the affected side before the pleural fluid is obtained.
* Medical or psychological impediment to probable compliance with the protocol.
* Patients on steroid (or other immunosuppressive agents) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation and must stop of any such treatment during the time of the study.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, superficial or in-situ cancer of the bladder or other cancer for which the patient has been disease-free for five years.
* Serious concomitant disease, no active infections. Patients with a history of autoimmune disease or organ allografts, or with active acute or chronic infection, including HIV (as determined by ELISA and confirmed by Western Blot) and viral hepatitis (as determined by HBsAg and Hepatitis C serology).
* Patients with serious intercurrent chronic or acute illness such as pulmonary (asthma or COPD) or cardiac (NYHA class III or IV) or hepatic disease or other illness considered by the study coordinator to constitute an unwarranted high risk for investigational DC treatment.
* Patients with a known allergy to shell fish (may contain KLH).
* Pregnant or lactating women.
* Patients with inadequate peripheral vein access to perform leukapheresis
* Concomitant participation in another clinical trial
* An organic brain syndrome or other significant psychiatric abnormality which would comprise the ability to give informed consent, and preclude participation in the full protocol and follow-up.
* Absence of assurance of compliance with the protocol. Lack of availability for follow-up assessment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
number of cytotoxic T cells and regulatory T cells in the blood of patients | up to 1 year
  2 weeks before, inbetween (2-weekly, 3 times) and 2 weeks after DC treatment, 7 ml blood samples are collected.

SECONDARY OUTCOMES:
safety and toxicity | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Aerts, PhD MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Hegmans JP, Hemmes A, Aerts JG, Hoogsteden HC, Lambrecht BN. Immunotherapy of murine malignant mesothelioma using tumor lysate-pulsed dendritic cells. Am J Respir Crit Care Med. 2005 May 15;171(10):1168-77. doi: 10.1164/rccm.200501-057OC. Epub 2005 Mar 11. PMID 15764728
- [Background] Hegmans JP, Veltman JD, Lambers ME, de Vries IJ, Figdor CG, Hendriks RW, Hoogsteden HC, Lambrecht BN, Aerts JG. Consolidative dendritic cell-based immunotherapy elicits cytotoxicity against malignant mesothelioma. Am J Respir Crit Care Med. 2010 Jun 15;181(12):1383-90. doi: 10.1164/rccm.200909-1465OC. Epub 2010 Feb 18. PMID 20167848
- [Background] Veltman JD, Lambers ME, van Nimwegen M, de Jong S, Hendriks RW, Hoogsteden HC, Aerts JG, Hegmans JP. Low-dose cyclophosphamide synergizes with dendritic cell-based immunotherapy in antitumor activity. J Biomed Biotechnol. 2010;2010:798467. doi: 10.1155/2010/798467. Epub 2010 May 23. PMID 20508851
- [Derived] van Gulijk M, Belderbos B, Dumoulin D, Cornelissen R, Bezemer K, Klaase L, Dammeijer F, Aerts J. Combination of PD-1/PD-L1 checkpoint inhibition and dendritic cell therapy in mice models and in patients with mesothelioma. Int J Cancer. 2023 Apr 1;152(7):1438-1443. doi: 10.1002/ijc.34293. Epub 2022 Oct 3. PMID 36104949
- [Derived] Cornelissen R, Hegmans JP, Maat AP, Kaijen-Lambers ME, Bezemer K, Hendriks RW, Hoogsteden HC, Aerts JG. Extended Tumor Control after Dendritic Cell Vaccination with Low-Dose Cyclophosphamide as Adjuvant Treatment in Patients with Malignant Pleural Mesothelioma. Am J Respir Crit Care Med. 2016 May 1;193(9):1023-31. doi: 10.1164/rccm.201508-1573OC. PMID 26652184